CLINICAL TRIAL: NCT07105917
Title: Sodium-dependent Glucose Transporters 2 Inhibitor for Neuroprotection in Patients With Acute Ischemic Stroke
Brief Title: SLGT2i for Neuroprotection in Patients With Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Min Lou, Principal Investigator, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNPS
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: SGLT2i with standard therapy (Experimental): Any of the following SGLT2 inhibitors (SGLT2i) can be selected for treatment:
  Dapagliflozin 10 mg once daily (QD) or Empagliflozin 10 mg once daily (QD) If the patient has concurrent diabetes, the use of other antidiabetic drugs is not restricted.
  The treatment should last for at least 14 days.
  Interventions: Drug: SGLT-2 inhibitors
- Standard therapy (Sham Comparator): According to the guideline-recommended standard treatment, if the patient has diabetes, there is no restriction on the use of other antidiabetic drugs (except SGLT-2 inhibitors).
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Drug: SGLT-2 inhibitors — Any of the following SGLT2 inhibitors (SGLT2i) can be selected for treatment:
  Dapagliflozin 10 mg once daily (QD) or Empagliflozin 10 mg once daily (QD) If the patient has concurrent diabetes, the use of other antidiabetic drugs is not restricted.
  The treatment should last for at least 14 days.
  Arms: Experimental: SGLT2i with standard therapy
Other: Standard medical treatment — According to the guideline-recommended standard treatment, if the patient has diabetes, there is no restriction on the use of other antidiabetic drugs (except SGLT-2 inhibitors).
  Arms: Standard therapy

SUMMARY:
Stroke is a leading cause of disability and mortality globally. With population aging, ischemic stroke (80% of cases) has become China's primary cause of adult disability. Sodium-dependent glucose transporters 2 inhibitors （SGLT2i） demonstrate cardiovascular protection beyond glycemic control, even in patients without diabetes.

Preclinical studies suggest neuroprotective effects via improving cerebral glucose metabolism, anti-inflammatory/antioxidant actions, and reducing neuronal apoptosis. Therefore, the investigators aim to evaluate whether SGLT2i could improve 3-month functional outcomes (mRS scores) in AIS patients compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with acute ischemic stroke (AIS) within ≤ 3 days of onset, with no restrictions on reperfusion therapy
* NIHSS score of 4-25 at the time of randomization
* Pre-stroke mRS score ≤ 1
* Signed informed consent form

Exclusion Criteria:

* Presence of intracranial hemorrhage at the time of randomization
* BMI ≤ 18 kg/m²
* Severe renal insufficiency (eGFR < 30 mL/min) or severe liver impairment (Child-Pugh Class C liver function)
* Type 1 diabetes mellitus
* Blood glucose level < 2.7 mmol/L or > 22.2 mmol/L at the time of randomization
* Systolic blood pressure < 95 mmHg at the time of randomization
* History of heart failure
* Use of SGLT-2 inhibitors within 4 weeks prior to randomization
* Intolerance to SGLT-2 inhibitors
* Life expectancy < 3 months
* Pregnant or lactating women
* Already enrolled in another clinical trial
* Other conditions deemed inappropriate for inclusion by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of mRS scores at 3 months | 3 months

SECONDARY OUTCOMES:
Proportion of patients with mRS scores 0-1 at 3 months | 90 days
Proportion of patients with mRS scores 0-2 at 3 months | 90 days
Proportion of patients with mRS scores 0-3 at 3 months | 90 days
NIHSS scores at Day 7 post-onset/at discharge | 7 days
Change in NIHSS scores from randomization to Day 7 post-onset/at discharge | 7 days
All-cause mortality | 90 days
Stroke-related mortality | 90 days
Symptomatic intracranial hemorrhage within 14 days | 14 days
Early neurological deterioration, defined as an increase of ≥4 points in NIHSS scores from randomization to Day 7 post-onset/at discharge | 7 days
Serious adverse events within 3 months | 90 days
Adverse events leading to discontinuation of SGLT2i | 14 days
Adverse events related to SGLT2i (volume depletion, renal events, severe hypoglycemic events, fractures, diabetic ketoacidosis, amputations) | 90 days